CLINICAL TRIAL: NCT03497962
Title: Using P4 Peptide to Augment Ex Vivo Phagocyte Function in Patients with Severe Community Acquired Pneumonia (CAP)
Brief Title: P4 Peptide in Community Acquired Pneumonia
Acronym: P4
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 12/NW/0730
Record Dates: First submitted 2015-05-08; First posted 2018-04-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2017-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Blood Specimen Collection; Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
  bronchoalveolar lavage (BAL)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ITU patients: 25 patients will be recruited from the Intensive Care Unit/ High dependency unit Inclusion- Adults (>18years) with community acquired pneumonia (CAP).
  Interventions: Procedure: Venepuncture; Procedure: Bronchoscopy
- Healthy volunteer: 24 healthy adult volunteers will be recruited to establish a comparison data set and to extend the laboratory observations to include other bacterial pathogens.
  Interventions: Procedure: Venepuncture; Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Venepuncture — Taken from established arterial or central lines in critical care setting or by experienced clinicians if no line available and in healthy volunteers.
Procedure: Bronchoscopy — Broncho-alveolar lavage to obtain alveolar macrophages

SUMMARY:
The investigators' aim is to find out whether immune cells from patients with a severe chest infection will react ex vivo to a new immunomodulating peptide, P4 as part of augmented passive immunotherapy

The investigators know that P4 treatment can successfully improve the efficiency of specialized immune cells responsible for killing bacteria. The investigators also know that P4 treatment is effective in healthy human volunteers but wish to extend this observation to patients that have infection, as immune cells may react differently in these patients. If this study is successful, the investigators hope to be moving closer to a new treatment against severe bacterial infections.

The investigators plan to recruit patients admitted to the Intensive Care Unit (ICU) and healthy volunteers, using carefully established inclusion and exclusions criteria with severe community acquired pneumonia (CAP) and obtain both blood and (if clinically feasible), a bronchoscopy BAL sample (washing of lung tissue).

DETAILED DESCRIPTION:
The investigators will examine the response to P4 peptide of alveolar macrophages from bronchoalveolar lavage (BAL) and neutrophils from peripheral blood collected from patients with severe pneumonia admitted to the ITU.

The investigators expect to show improved phagocytosis, oxidative burst, cellular activation (flow cytometry, electron microscopy, cytokine production, transcriptomics) and bacterial killing when P4 is used to stimulate immune cells and this may lead to a novel approach to the treatment of severe infections.

The investigators will also examine the effect of P4 on alveolar macrophages and neutrophils from healthy volunteers in order to ensure comparability with previously published results and extend observations using S.pneumoniae to other causes of severe pneumonia including E.coli, Salmonellae, M.tuberculosis and Pseudomonas.

Augmented passive immunotherapy (API) is a novel potential treatment strategy to combat fulminant bacterial infections. It consists of two components

1. a peptide that enhances bacterial uptake and killing by phagocytes.
2. exogenous antibody (provided with intravenous immunoglobulin, a licensed medicinal product) which optimizes the phagocytosis. Previous studies of API have included extensive murine studies of acute and chronic bacterial infection with several different organisms. P4 has also been tested in aged mice and in mucosal administration.

The investigators will recruit patients with severe community acquired pneumonia on ICU and healthy volunteers using carefully established inclusion and exclusions criteria.

This research seeks to establish proof-of-concept for augmented passive immunotherapy in patients with severe pneumonia. Patients with mild to moderate pneumonia often respond to antibiotic therapy but those with severe community-acquired pneumonia who require admission to Intensive Care have a hospital mortality of 49.4%, despite antibiotics and optimal supportive care. These patients represent 6% of all admissions to Intensive Care Units in the UK. Strategies to improve clinical outcome for this group of patients are much needed and the investigators' research cohort has been selected to represent this group. The immunological characteristics of patients with overwhelming sepsis are likely to differ from patients with milder infection. Immune cells taken from patients with milder forms of sepsis may not respond to in vitro stimulation in the same way as cells taken from severely septic patients and therefore should not be used to establish proof-of-concept for a therapy intended for critically ill patients on Intensive Care.

ELIGIBILITY:
Inclusion Criteria for ITU patients:

* Adults (>18y) with community acquired pneumonia.
* Diagnosis of CAP upon hospital admission requires: Radiographic shadowing unexplained by other causes plus Symptoms/signs consistent with acute lower respiratory tract infection.

Exclusion Criteria for ITU patients:

* Previous hospital admission within 14 days (implies hospital acquired).
* Immunocompromising comorbidity or therapy (e.g. HIV infection, chemotherapy).
* Pregnancy.
* Deemed inappropriate by responsible Intensivist. Already recruited in to an interventional study (where the study therapy may influence the results of this study).
* Failure to obtain consent.

Bronchoscopy Exclusion criteria (ITU patients):

* The patient does not require a bronchoscopy for clinical reasons
* The patient is not invasively ventilated therefore not requiring a bronchoscopy
* The patient condition deteriorates prior to bronchoscopy such that they might no longer tolerate the procedure (e.g. those progressing to require high frequency oscillation, prone-positioning, PEEP>15cmH2O or FiO2>0.8 for ventilation).
* Patient does not tolerate bronchoscopy, i.e. if there is oxygen desaturation to <90% for >60 seconds or haemodynamic disturbance during the procedure.
* The intensive care clinician responsible for the patient develops any new concerns about the safety of bronchoscopy or bronchoalveolar lavage.

Inclusion/ Exclusion Criteria for healthy volunteers:

* Adults (>18y).
* Able to give fully informed consent.
* Fluent English speaker.
* Non-smoking.
* Healthy adults without current illness.
* Contraindication to bronchoscopy or immunomodulatory medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted into the intensive care unit with community aquired pneumonia (CAP)
  Healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Number of bacteria phagocytosed from neutrophils and macrophages stimulated with P4 compared to unstimulated cells.comparing cells stimulated with P4 and unstimulated cells. | 12 hours
  Opsonophagocytic killing assay performed on blood neutrophils and BAL macrophages. Neutrophils and macrophages are stimulated with P4, control is unstilumated neutrophils and macrophages. The comparison is made between the killing of pneumococcal bacteria between the stimulated and unstimulated cells.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Gordon, Professor, Principal Investigator — Royal Liverpool University Hospital/ Liverpool School of Tropical Medicine
Locations (1):
- Royal Liverpool University Hospital, Liverpool, Merseyside, United Kingdom